CLINICAL TRIAL: NCT06741397
Title: A Phase 2b Single Arm, Repeat Dose Study to Evaluate the Pharmacokinetic Profile, Safety, and Tolerability of A New Formulation of Cabotegravir LA Injected Intramuscularly Q4M in Adolescent and Adult Participants at Risk of HIV Acquisition
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of a New Formulation of Cabotegravir Long-Acting Administered Intramuscularly in a 4-month Dosing Interval (Q4M)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 219230; 2024-000061-24 (EudraCT Number)
Record Dates: First submitted 2024-12-17; First posted 2024-12-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: HIV Infections
Keywords: Cabotegravir (CAB); New formulation of CAB LA; CAB LA; HIV; 4-month dosing interval (Q4M); Safety
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Masking Description: This is an open label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CAB Group (Experimental): Participants receive lead-in injections comprising cabotegravir LA during month one and injections of a new formulation of CAB LA at Month 3, Month 5 and every 4 months thereafter to Month 29.
  Interventions: Drug: CAB LA; Drug: New formulation of CAB LA

INTERVENTIONS:
Drug: CAB LA — Injections administered IM gluteal.
Drug: New formulation of CAB LA — Injections administered IM gluteal.

SUMMARY:
This study will evaluate the pharmacokinetics (PK), safety, and tolerability of a new formulation of Cabotegravir (CAB) dosed every 4-months (Q4M) for pre-exposure prophylaxis (PrEP) in participants at risk of HIV-1 acquisition.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of obtaining informed consent, adolescent and adult participants weighing at least 35 kg.
2. Participants must have a nonreactive HIV test at Screening (rapid test, nonrapid HIV immunoassay, and HIV RNA) and enrollment (a rapid test, nonrapid HIV immunoassay, and HIV RNA).
3. Participants who are at risk of acquiring HIV, defined as having had anal or vaginal sex in the past 6 months.
4. Participants who are overtly healthy as determined by medical evaluation by a responsible and experienced physician, including medical history, physical examination, laboratory tests and cardiac monitoring at the time of screening.
5. No alcohol or substance use that, in the opinion of the study investigator and medical monitor, would interfere with the conduct of the study (e.g., provided by self-report, or found upon medical history and examination or in available medical records).
6. Participants who have received oral PrEP are eligible, but they must discontinue oral PrEP within 10 days of Day 1 visit.
7. Male or female at birth, (transgender individuals are not excluded). Contraceptive use should align with local regulations. Participants assigned female at birth must not be pregnant or breastfeeding and must either not be of childbearing potential (POCBP) or use highly effective contraception. A POCBP must have a negative pregnancy test within 30 days before dosing.
8. Participants must be >=16 years old, of legal age to consent to sexual intercourse, and capable of giving written informed consent. Adolescents must provide written informed assent/consent and/or obtain parental/guardian consent if not of legal age, as per site SOPs and IRB/EC policies.

Exclusion Criteria:

1. One or more reactive or positive HIV test results at Screening or Enrollment, even if HIV infection was not confirmed.
2. Participants who are breastfeeding or plan to become pregnant or breastfeed during the study.
3. Alanine aminotransferase (ALT) >=3 times the upper limit of normal (ULN).
4. Evidence of active Hepatitis B virus (HBV) infection.

   * Participants positive for HBsAg or HBV DNA are excluded.
   * Participants negative for anti-HBs but positive for anti-HBc (negative HBsAg status) and positive for HBV DNA are excluded.
5. Unstable liver disease, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
6. History of clinically relevant hepatitis within last 6 months.
7. Known history of liver cirrhosis with or without viral hepatitis co-infection.
8. Participants with Hepatitis C virus (HCV) co-infection will be allowed entry into this study if:

   * Liver enzymes meet entry criteria.
   * HCV Disease has undergone appropriate work-up, and is not advanced, and will not require treatment prior to the primary endpoint (e.g., Month 13).
   * In the event that recent biopsy or imaging data is not available or inconclusive, the Fibrosis 4 (Fib-4) score will be used to verify eligibility:

     i. Fib-4 score greater than (>) 3.25 is exclusionary. ii. Fib-4 scores 1.45 - 3.25 requires Medical Monitor consultation. Fibrosis 4 score Formula: (Age x AST) / (Platelets x (sqr [ ALT]) It is approved by the Medical Monitor.
9. Estimated glomerular filtration rate of <30 mL/min/1.73 m^2 via CKD-EPIcr_R (2021) method.
10. Any acute laboratory abnormality at Screening, which, in the opinion of the investigator, would preclude the participant's participation in the study of an investigational compound.
11. Any verified Grade 4 laboratory abnormality, with the exception of Grade 4 [triglycerides or lipid abnormalities].
12. Participants determined by the Investigator to have a high risk of seizures, A participant with a prior history of seizure may be considered for enrolment if the Investigator believes the risk of seizure recurrence is low. All cases of prior seizure history should be discussed with the Medical Monitor prior to enrolment.
13. Participant is currently participating in or has participated in a study with a compound or device that is not commercially available within 30 days of signing informed consent, unless permission from the Medical Monitor is granted.
14. Presence of any history of allergy/sensitivity to any of the study drug.
15. Inflammatory skin conditions that compromise the safety of IM injections, per the discretion of the investigator.
16. Participant has an implant/enhancement (including fillers) at the area of proposed injection (e.g., gluteus medius); or tattoo or other dermatological condition overlying the area for IM (e.g., gluteus medius) or any other area which may significantly interfere with interpretation of injection site reactions.
17. Current or anticipated need for chronic anti-coagulants or active coagulopathy (primary or iatrogenic) which would contraindicate IM injection.
18. Ongoing or clinically relevant pancreatitis.
19. Clinically significant cardiovascular disease or history of clinically significant cardiovascular disease.
20. All participants will be screened for STIs (e.g., chlamydia, gonorrhea, trichomoniasis, syphilis). Participants with untreated infections are excluded. Participants may be rescreened at least 24 hours after completion of STI treatment.
21. History or presence of sensitivity to any of the study medications or their components or drugs of their class, or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation. In addition, if heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
22. Ongoing uncontrolled malignancy is excluded, whereas participants who have controlled localized malignancies may be included on agreement between the investigator and the Medical Monitor.
23. Participants who in the investigator's judgment, poses a significant suicidality risk.
24. Any pre-existing physical or mental condition (including substance abuse disorder) which, in the opinion of the Investigator or the medical monitor, may interfere with the participant's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the participant.
25. Any condition which, in the opinion of the Investigator or the medical monitor, may interfere with the absorption, distribution, metabolism or excretion of the study drugs or render the participant unable to receive IM medication.
26. Co-enrollment in any other interventional research study or other concurrent studies which may have interfered with this study (as provided by self-report or other available documentation). Exceptions for non-interventional studies may be made if appropriate after consultation with the Medical Monitor.
27. Participants receiving any protocol-prohibited medication and who are unwilling or unable to switch to an alternate medication.
28. Use of antiretroviral therapy (ART) for Postexposure Prophylaxis within the 90 days prior to Day 1.
29. Use of CAB LA for PrEP at any time prior to Screening.
30. Exposure to an experimental drug or experimental vaccine within either 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of IP.
31. Anticipated need for HCV therapy with interferon or any drugs that have potential for adverse drug:drug interactions with study treatment throughout the entire study period.
32. Treatment with an HIV-1 preventive vaccine within 90 days of Screening.
33. Participant is unlikely to adhere to the study procedures, keep appointments, is planning to relocate during the study, or remain on study through to its conclusion.
34. Participants who are considered high-risk, meeting at least one of the following criteria:

    * Participant who has exchanged condomless sex for goods or money within the past 12 months prior to Screening.
    * Participant who has used recreational intravenous drugs within the past 12 months prior to Screening.
    * Participant who has participated in Chemsex practice (such as the use of cocaine, crack cocaine, methamphetamine, ketamine, 3,4-methlenedioxy-methamphetamine, GHB, mephedrone or prescription drugs apart from those prescribed by a licensed provider) within the past 6 months prior to Screening.
    * Participant with any STI in the last 6 months also reporting any partners for condomless sex.
    * Participant who has condomless sex with a serodiscordant partner who has a detectable viral load or is not on ART.
    * Participant with any other behavior assessed by the investigator as high-risk sexual behavior.
35. Participant has in the last 14 days prior to Screening presented with signs and symptoms, which, in the opinion of the investigator, are suggestive of acute HIV infection. Participants may only be enrolled if clinical suspicion of HIV is ruled out with non-reactive results.
36. Participant becomes a ward of state (e.g., child in care).

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-09-09 (Estimated); Study Completion 2029-01-10 (Estimated)

PRIMARY OUTCOMES:
CAB trough concentrations for target of 1.05 microgram per milliliter (μg/mL) for men and 1.39 μg/mL for women | From Month 13 to Month 25
  CAB trough concentrations are evaluated at or above the target of 1.05 μg/mL for men and 1.39 μg/mL for women, once steady state has been achieved, but no earlier than Month 13 of the study.

SECONDARY OUTCOMES:
CAB trough concentrations for target of 0.672 μg/mL for men and 0.683 μg/mL for women | At Month 1
  CAB trough concentrations are evaluated at or above the target of 0.672 μg/mL for men and 0.683 μg/mL for women.
CAB trough concentrations for target of 1.05 μg/mL for men and 1.39 μg/mL for women following loading dose | From Month 3 to Month 33
  CAB trough concentrations are evaluated at or above the target of 1.05 μg/mL for men and 1.39 μg/mL for women.
CAB plasma concentrations | At Day 1, Day 1+1Week (W), Month (M) 1, M1+1W, M2, M3, M3+1W, M4, M5, M5+1W, M6, M7, M8, M9, M9+1W, M10, M11, M13, M13+1W, M17, M17+1W, M21, M25, M29, and M33
  Blood samples are collected by visit.
CAB trough concentrations for target of 4x PA-IC90 | At Months 1, 3, 5, 9, 13, 17, 21, 25, 29, and 33
  CAB trough concentrations are evaluated at or above the target of 4 times (4x) PA-IC90. PA-IC90 is defined as protein-adjusted concentration at which 90% inhibition of viral replication is achieved.
Percentage of participants with confirmed incident HIV infections | Up to Month 33
Percentage of participants with Study Medication Satisfaction Questionnaire Status version (SMSQs) results | From Month 1 up to Month 33
  SMSQs is a self-completion measure which is evaluating 11-items (i.e., satisfaction, side effects, demands, convenience, flexibility, understanding, lifestyle, recommend, continue, easy or difficult, discomfort or pain). SMSQs is self-administered at each planned study visit and prior to the study drug administration.
Percentage of participants with Adverse events (AEs) | Up to Month 33
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment.
Percentage of participants with AEs by severity | Up to Month 33
  Severity is graded according to the Division of Acquired Immunodeficiency Syndrome (DAIDS) grading criteria, where Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = potentially life-threatening.
Percentage of participants with laboratory abnormalities | Up to Month 33
Percentage of participants with laboratory abnormalities by severity | Up to Month 33
  Severity is graded according to the DAIDS grading criteria, where Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = potentially life-threatening.
Percentage of participants with changes in laboratory parameters | Up to Month 33

CONTACTS AND LOCATIONS:
Locations (23):
- United States (22):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Palm Springs, California
  - GSK Investigational Site, Doral, Florida
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Berkley, Michigan
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Valhalla, New York
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Seattle, Washington
- GSK Investigational Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Study sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf